CLINICAL TRIAL: NCT01878331
Title: Long-term, Prospective, Cohort Study to Evaluate Safety and Efficacy of Two Different Dental Implant Alloys in Straumann 3.3mm Diameter Bone Level Implants for Removable Prosthesis in Patients With Edentulous Mandibles
Brief Title: Long-term Study to Evaluate Different Dental Implant Alloys in Straumann 3.3mm Diameter Bone Level Implants
Status: Completed | Type: Observational
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR 01/13
Record Dates: First submitted 2013-04-29; First posted 2013-06-14 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Jaw, Edentulous
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Roxolid: Patient do not receive an intervention in the extension study. Rather they are followed on the implant treatment from the core study which included a split-mouth design where all patients received both a Roxolid and SLActive implant.
- SLActive: Patient do not receive an intervention in the extension study. Rather they are followed on the implant treatment from the core study which included a split-mouth design where all patients received both a Roxolid and SLActive implant.

SUMMARY:
Patients with an edentulous mandible restored with implants who have participated in the core study CR 04/07 will be recruited for this extension study. No further interventions will be made for this extension study other than a clinical follow-up examination and questionnaires. Patients will not receive an investigational treatment in this study. Patients will be followed at 5 to 10 years from the date of the original implant loading

DETAILED DESCRIPTION:
The primary study objective is to compare implant survival with the Titanium Zirconium (Roxolid™) implant compared the Titanium grade IV (SLActive®) implant between baseline (surgery) and 10 years.

The following outcome parameters will be evaluated at 5 and 10 years post surgery for the two different implant types Straumann® Bone Level SLActive, diameter 3.3 mm, Titanium-Zirconium (Roxolid®) vs. Straumann® Bone Level SLActive implant, diameter 3.3 mm, Titanium Grade IV:

* Implant survival
* Implant success according to Buser et al. (1990)
* Crestal bone level change measured by Orthopantomogram (OPT)
* Soft tissue health
* Clinical measurements
* Prosthetic parts assessments: Success and maintenance
* Oral Health Related Quality of Life (OHRQoL)
* Product Safety (Adverse events and device deficiencies)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form
* Patients must be committed to participate in the study until the ten year follow-up examinations
* Subjects must have received treatment in the CR 04/07 core study
* Subjects must have completed 3 year visit of core study

Exclusion Criteria:

* Physical handicaps that would interfere with the ability to perform adequate oral hygiene or attend follow up visits
* Use of any investigational drug or device during the study
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patient ≥ 18 years of age who were provided with an implant supported over-denture in the mandible in the course of the core study (CR 04/07).
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Implant Survival | 10 years following implant procedure date
  This is a long term follow up extension study including evaluations at 5 and 10 years after the implant procedure from the core study. Implant survival will be assessed based on surviving implants for all patients at 10 years.

SECONDARY OUTCOMES:
Crestal bone level change | 5 and 10 years
  The change in crestal bone level will be measured on standard x-rays taken at 5 and 10 years as per standard of care. An independent reviewer will evaluate all x-rays for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Frauke Müller, Prof., Study Chair — University of Geneva; Bilal Al-Nawas, Prof., Principal Investigator — Klinikum der Johannes - Gutenberg - Universität Mainz; Eugenio Romeo, Prof., Principal Investigator — Università degli Studi di Milano, Dipartimento di Medicina, Chirurgia e Odontoiatria; Joke Duyck, Prof., Principal Investigator — Department of Oral Health Sciences, Catholic University (KU) Leuven; Torsten E Reichert, Prof., Principal Investigator — Klinikum der Universität Regensburg; Alessandro Perucchi, Prof., Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Frauke Müller, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller F, Al-Nawas B, Storelli S, Quirynen M, Hicklin S, Castro-Laza J, Bassetti M, Srinivasan M; Roxolid Study Group. Small-diameter titanium grade IV and titanium-zirconium implants in edentulous mandibles: Ten-year results from a double-blind, randomised controlled split-mouth core-trial. Clin Oral Implants Res. 2024 Jan;35(1):77-88. doi: 10.1111/clr.14199. Epub 2023 Nov 9. PMID 37942666
- [Derived] Muller F, Al-Nawas B, Storelli S, Quirynen M, Hicklin S, Castro-Laza J, Bassetti R, Schimmel M; Roxolid Study Group. Small-diameter titanium grade IV and titanium-zirconium implants in edentulous mandibles: five-year results from a double-blind, randomized controlled trial. BMC Oral Health. 2015 Oct 12;15(1):123. doi: 10.1186/s12903-015-0107-6. PMID 26458813